CLINICAL TRIAL: NCT02483611
Title: Effect of Intravenous Infusion of Magnesium Sulfate Associated or Not to Lidocaine On the Neuromuscular Blockade Induced by Muscle Relaxant Cistracurium
Brief Title: Effects of Intravenous Lidocaine Associated With Magnesium Sulfate on the Cisatracurium-Induced Neuromuscular Block
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Waynice N.P. Garcia, M.D., Ph.D, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: 5362/2013; 15541213.3.0000.5440 (Registry Identifier: [Plataforma Brasil])
Record Dates: First submitted 2015-06-18; First posted 2015-06-29 (Estimated); Results first posted 2016-01-15 (Estimated); Last update posted 2016-01-15 (Estimated); Status verified 2015-12

CONDITIONS: Neuromuscular Block
Keywords: Onset; Recovery; Lidocaine; Cisatracurium; Magnesium sulfate; Isotonic solution
MeSH Terms: interventions — Magnesium Sulfate; Lidocaine; Isotonic Solutions; cisatracurium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group M (Experimental): Magnesium Sulfate. In this group, the patients received magnesium sulfate 40 mg/Kg as a bolus and 20 mg/kg/h by continuous IV infusion during surgery.
  After the bolus of magnesium sulfate, 0.15 mg/kg of cisatracurium was infused over 5 seconds.
  Interventions: Drug: Magnesium Sulfate; Drug: Cisatracurium
- Group ML (Experimental): Magnesium Sulfate plus Lidocaine. In this group, the patients received 40 mg/kg of Magnesium Sulfate plus 3 mg kg-1 lidocaine as a bolus and 20 mg/kg/h and 3 mg/kg/h, respectively, by infusion continuously during the surgery.
  After the bolus of magnesium sulfate and lidocaine, 0.15 mg/kg of cisatracurium was infused over 5 seconds
  Interventions: Drug: Magnesium Sulfate; Drug: Lidocaine; Drug: Cisatracurium
- Group C (Placebo Comparator): Isotonic Solution. In this group, the patients received the volume of isotonic solution equivalent to the volume of solution infused into experimental groups.
  After the bolus of the isotonic solution , 0.15 mg/kg of cisatracurium was infused over 5 seconds
  Interventions: Drug: Isotonic Solution; Drug: Cisatracurium

INTERVENTIONS:
Drug: Magnesium Sulfate
  Arms: Group M; Group ML
Drug: Lidocaine
  Arms: Group ML
Drug: Isotonic Solution
  Arms: Group C
Drug: Cisatracurium
  Other Names: Nimbex

SUMMARY:
The magnesium sulfate and lidocaine have been increasingly used alone or in combination during anesthesia procedure to meet various objectives, such as reduction of pain, use of smaller anesthetic doses and stabilization of hemodynamic parameters.

These medicines are often used in combination with neuromuscular blocking agents, which may contribute to the occurrence of residual block in some patients after anesthetic procedures. It was estimated that only 1-3 % of patients with residual block developing clinically apparent events. In a small proportion of patients, the consequences of residual blockade are very serious and even lethal. It is estimated that 40 % of patients with muscle paralysis come to the post-anesthesia care unit (PACU).

Considering that: (a) magnesium sulfate and lidocaine are showing an increasing number of applications in various areas of medicine, (b) these medications stand out for their properties analgesic, anti-inflammatory, anti-arrhythmic, neuroprotective and capable of reducing the demand of anesthetics and opioids, (c) magnesium sulfate as lidocaine has been important part of the therapeutic arsenal to control a large number of diseases (d) the patient surgical surgery or potentially have benefited in particular from its effects, (and) these drugs have been used routinely in many medical services as well as adjuvants in anesthesia, (f) previous studies have shown that magnesium sulfate is able to prolong the duration of neuromuscular blockade by different types of muscle relaxants, with controversies about its effect on latency (g) the effect of lidocaine on the action of muscle relaxants in current literature have shown great controversy and (h) do not exist in the literature studies involving both drugs; the investigators aimed to investigate the effects of magnesium sulphate infused alone or associated with lidocaine on the neuromuscular blockade promoted by cisatracurium, as well as evaluate its possible hemodynamic repercussions. For this purpose the SM was infused in bolus, prior to tracheal intubation and continuously during the maintenance of general anesthesia; the Lidocaine, when associated and the Isotonic Solution were used in the same way and timeline as SM. As secondary objectives it has been proposed to evaluate if the Lidocaine with Magnesium Sulfate would be able to interfere with the hemodynamic stability of the patients in the study.

DETAILED DESCRIPTION:
The study was approved by the Medical Research Ethics Committee of the Hospital das Clinicas, of the Faculty of Medicine of Ribeirao Preto, University of Sao Paulo, Brazil; Its Unique Protocol ID is 5362/2013. This study was conducted with free written informed consent from the study subjects.

This report describes a prospective randomized clinical trial. The author states that the report includes every item in the checklist for a prospective randomized clinical trial.

The study was registered prior to patient enrollment. Forty-eight American Society of Anesthesiology patient classification status ASA I and II undergoing elective surgery were divided into three parallel groups. The M group received MS 40 mg.kg-1 as a bolus before the induction of anesthesia and 20mg.kg-1h-1 via continuous i.v. infusion during the operation period. The ML group received identical doses of MS combined with lidocaine 3 mg.kg-1 as a bolus before the induction of anesthesia and 3 mg.kg-1h-1 via continuous i.v. infusion during the operation period. The control group was administered a equivalent volume of isotonic solution. Anesthesia was maintained via propofol and remifentanil infusions. After loss of patient consciousness and administration of the bolus infusions, a 0.15 mg.kg-1 bolus of cisatracurium was administered to the patient over 5 s. No additional cisatracurium injections were performed. The patient's neuromuscular function was assessed every 15 s by measuring the adductor polis with a TOF Watch SX acceleromyograph. The primary endpoint was the time at which spontaneous recovery of a train-of-four (TOF) ratio of 90% as achieved. The systolic, diastolic and mean and heart rate were recorded and annotated at various times: M1- when the patient arrived in the operating room; M2- immediately before induction of anesthesia; M3- before the infusion of the tested solutions (saline, magnesium sulphate or magnesium sulphate associated with lidocaine); M4- five minutes after M3 (end of infusion loading dose of test solutions); M5 immediately before intubation; M6- one minute after tracheal intubation and M7 (a through f) - every fifteen minutes until the end of the study.

The sample size was calculated with a power of 80% to detect differences of 20% in the timing of clinical onset and the duration of the neuromuscular blockade (NMB). Quantitative variables were described as mean ± standard deviation. The normality of the distributions was tested for all variables in each group, using the non-parametric test of Shapiro-Wilk. When the variable normally distributed, we used the analysis of variance test (ANOVA) for comparison between groups. When differences were found between the groups, we used the Tukey test for multiple comparisons. When the variable is not normally distributed by applying the Shapiro-Wilk test, we used the Kruskal-Wallis test to compare the groups. When differences were found between the groups, we used the Dunn test for multiple comparisons. The critical level of significance was 5%.

During the analysis of the recovery characteristics of the neuromuscular blockade, all parameters based on the T1 response (DUR 25% DUR 75% and DUR 95%) were normalized considering the final T1 value when this response did not return to baseline (VIBY-MOGENSEN et al., 1996).

ELIGIBILITY:
Before the recruitment of patients, the study was approved by Brazil Platform (a national and unified basis of research involving human subjects records) and published by the ClinicalTrials.gov

Inclusion Criteria:

* ASA I or II
* BMI between 18 and 29

Exclusion Criteria:

* Use of medications that could affect the neuromuscular blockade such as calcium channel inhibitors, anticonvulsants and lithium carbonate
* Presence of neuromuscular, renal or hepatic dysfunction.
* Hypermetabolic or hypometabolic states such as fever, infection, and hyperthyroidism or hypothyroidism
* Acid-base disorder, congestive heart failure or conductive heart problems, and those who were being treated for cardiac arrhythmias

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2015-07; Primary Completion 2015-08 (Actual); Study Completion 2015-09 (Actual)

REFERENCES:
- [Background] Murphy GS, Brull SJ. Residual neuromuscular block: lessons unlearned. Part I: definitions, incidence, and adverse physiologic effects of residual neuromuscular block. Anesth Analg. 2010 Jul;111(1):120-8. doi: 10.1213/ANE.0b013e3181da832d. Epub 2010 May 4. PMID 20442260
- [Background] Debaene B, Plaud B, Dilly MP, Donati F. Residual paralysis in the PACU after a single intubating dose of nondepolarizing muscle relaxant with an intermediate duration of action. Anesthesiology. 2003 May;98(5):1042-8. doi: 10.1097/00000542-200305000-00004. PMID 12717123
- [Background] Kim MH, Oh AY, Jeon YT, Hwang JW, Do SH. A randomised controlled trial comparing rocuronium priming, magnesium pre-treatment and a combination of the two methods. Anaesthesia. 2012 Jul;67(7):748-54. doi: 10.1111/j.1365-2044.2012.07102.x. Epub 2012 Mar 15. PMID 22420830
- [Background] Habe K, Kawasaki T, Sata T. [A case of prolongation of rocuronium neuromuscular blockade in a pregnant patient receiving magnesium]. Masui. 2014 Jul;63(7):817-9. Japanese. PMID 25098146
- [Background] Doig GS, Simpson F. Randomization and allocation concealment: a practical guide for researchers. J Crit Care. 2005 Jun;20(2):187-91; discussion 191-3. doi: 10.1016/j.jcrc.2005.04.005. PMID 16139163
- [Background] Hans GA, Defresne A, Ki B, Bonhomme V, Kaba A, Legrain C, Brichant JF, Hans PC. Effect of an intravenous infusion of lidocaine on cisatracurium-induced neuromuscular block duration: a randomized-controlled trial. Acta Anaesthesiol Scand. 2010 Nov;54(10):1192-6. doi: 10.1111/j.1399-6576.2010.02304.x. Epub 2010 Sep 14. PMID 20840515
- [Background] Kim MH, Oh AY, Han SH, Kim JH, Hwang JW, Jeon YT. The effect of magnesium sulphate on intubating condition for rapid-sequence intubation: a randomized controlled trial. J Clin Anesth. 2015 Nov;27(7):595-601. doi: 10.1016/j.jclinane.2015.07.002. Epub 2015 Aug 25. PMID 26315876
- [Background] Shahrami A, Assarzadegan F, Hatamabadi HR, Asgarzadeh M, Sarehbandi B, Asgarzadeh S. Comparison of therapeutic effects of magnesium sulfate vs. dexamethasone/metoclopramide on alleviating acute migraine headache. J Emerg Med. 2015 Jan;48(1):69-76. doi: 10.1016/j.jemermed.2014.06.055. Epub 2014 Sep 30. PMID 25278139
- [Background] Ventham NT, Kennedy ED, Brady RR, Paterson HM, Speake D, Foo I, Fearon KC. Efficacy of Intravenous Lidocaine for Postoperative Analgesia Following Laparoscopic Surgery: A Meta-Analysis. World J Surg. 2015 Sep;39(9):2220-34. doi: 10.1007/s00268-015-3105-6. PMID 26044546
- [Background] Govindarajan R, Shah A, Reddy VS, Parithivel V, Ravikumar S, Livingstone D. Improving the functionality of intra-operative nerve monitoring during thyroid surgery: is lidocaine an option? J Clin Med Res. 2015 Apr;7(4):282-5. doi: 10.14740/jocmr2025w. Epub 2015 Feb 9. PMID 25699129
- [Result] Czarnetzki C, Lysakowski C, Elia N, Tramer MR. Time course of rocuronium-induced neuromuscular block after pre-treatment with magnesium sulphate: a randomised study. Acta Anaesthesiol Scand. 2010 Mar;54(3):299-306. doi: 10.1111/j.1399-6576.2009.02160.x. Epub 2009 Nov 16. PMID 19919585
- [Result] Czarnetzki C, Lysakowski C, Elia N, Tramer MR. Intravenous lidocaine has no impact on rocuronium-induced neuromuscular block. Randomised study. Acta Anaesthesiol Scand. 2012 Apr;56(4):474-81. doi: 10.1111/j.1399-6576.2011.02625.x. Epub 2012 Jan 19. PMID 22260297
- [Result] Hans GA, Bosenge B, Bonhomme VL, Brichant JF, Venneman IM, Hans PC. Intravenous magnesium re-establishes neuromuscular block after spontaneous recovery from an intubating dose of rocuronium: a randomised controlled trial. Eur J Anaesthesiol. 2012 Feb;29(2):95-9. doi: 10.1097/EJA.0b013e32834e13a6. PMID 22183158
- [Result] Kim SH, So KY, Jung KT. Effect of magnesium sulfate pretreatment on onset and recovery characteristics of cisatracurium. Korean J Anesthesiol. 2012 Jun;62(6):518-23. doi: 10.4097/kjae.2012.62.6.518. Epub 2012 Jun 19. PMID 22778886
- [Result] Kussman B, Shorten G, Uppington J, Comunale ME. Administration of magnesium sulphate before rocuronium: effects on speed of onset and duration of neuromuscular block. Br J Anaesth. 1997 Jul;79(1):122-4. doi: 10.1093/bja/79.1.122. PMID 9301400
- [Result] Cardoso LS, Martins CR, Tardelli MA. Effects of intravenous lidocaine on the pharmacodynamics of rocuronium. Rev Bras Anestesiol. 2005 Aug;55(4):371-80. doi: 10.1590/s0034-70942005000400001. English, Portuguese. PMID 19468625
- [Result] Nonaka A, Sugawara T, Suzuki S, Masamune T, Kumazawa T. [Pretreatment with lidocaine accelerates onset of vecuronium-induced neuromuscular blockade]. Masui. 2002 Aug;51(8):880-3. Japanese. PMID 12229137
- [Result] Vivancos GG, Klamt JG, Garcia LV. Effects of 2 mg.kg(-)(1) of intravenous lidocaine on the latency of two different doses of rocuronium and on the hemodynamic response to orotracheal intubation. Rev Bras Anestesiol. 2011 Jan-Feb;61(1):1-12. doi: 10.1016/S0034-7094(11)70001-0. PMID 21334502
- [Result] Ghodraty MR, Saif AA, Kholdebarin AR, Rokhtabnak F, Pournajafian AR, Nikzad-Jamnani AR, Shah A, Nader ND. The effects of magnesium sulfate on neuromuscular blockade by cisatracurium during induction of anesthesia. J Anesth. 2012 Dec;26(6):858-63. doi: 10.1007/s00540-012-1439-x. Epub 2012 Jul 3. PMID 22752440
- [Result] Rotava P, Cavalcanti IL, Barrucand L, Vane LA, Vercosa N. Effects of magnesium sulphate on the pharmacodynamics of rocuronium in patients aged 60 years and older: A randomised trial. Eur J Anaesthesiol. 2013 Oct;30(10):599-604. doi: 10.1097/EJA.0b013e328361d342. PMID 23635996
- [Result] Gupta K, Vohra V, Sood J. The role of magnesium as an adjuvant during general anaesthesia. Anaesthesia. 2006 Nov;61(11):1058-63. doi: 10.1111/j.1365-2044.2006.04801.x. PMID 17042843
- [Result] McCoy EP, Connolly FM, Mirakhur RK, Loan PB, Paxton LD. Nondepolarizing neuromuscular blocking drugs and train-of-four fade. Can J Anaesth. 1995 Mar;42(3):213-6. doi: 10.1007/BF03010679. PMID 7743572
- [Result] Viby-Mogensen J, Jorgensen BC, Ording H. Residual curarization in the recovery room. Anesthesiology. 1979 Jun;50(6):539-41. doi: 10.1097/00000542-197906000-00014. No abstract available. PMID 156513
- [Result] Kopman AF, Kumar S, Klewicka MM, Neuman GG. The staircase phenomenon: implications for monitoring of neuromuscular transmission. Anesthesiology. 2001 Aug;95(2):403-7. doi: 10.1097/00000542-200108000-00023. PMID 11506113
- [Result] Staals LM, Driessen JJ, Van Egmond J, De Boer HD, Klimek M, Flockton EA, Snoeck MM. Train-of-four ratio recovery often precedes twitch recovery when neuromuscular block is reversed by sugammadex. Acta Anaesthesiol Scand. 2011 Jul;55(6):700-7. doi: 10.1111/j.1399-6576.2011.02448.x. Epub 2011 May 16. PMID 21574968
- [Result] Katz RL, Gissen AJ. Effects of intravenous and intra-arterial procaine and lidocaine on neuromuscular transmission in man. Acta Anaesthesiol Scand Suppl. 1969;36:103-13. doi: 10.1111/j.1399-6576.1969.tb00482.x. No abstract available. PMID 4315659
- [Result] Matsuo S, Rao DB, Chaudry I, Foldes FF. Interaction of muscle relaxants and local anesthetics at the neuromuscular junction. Anesth Analg. 1978 Sep-Oct;57(5):580-7. doi: 10.1213/00000539-197809000-00014. PMID 568429
- [Result] Toft P, Kirkegaard Nielsen H, Severinsen I, Helbo-Hansen HS. Effect of epidurally administered bupivacaine on atracurium-induced neuromuscular blockade. Acta Anaesthesiol Scand. 1990 Nov;34(8):649-52. doi: 10.1111/j.1399-6576.1990.tb03165.x. PMID 2275325
- [Result] Loyola YC, Braga Ade F, Poterio GM, Sousa SR, Fernandes SC, Braga FS. [Influence of lidocaine on the neuromuscular block produced by rocuronium: study in rat phrenic-diaphragmatic nerve preparation.]. Rev Bras Anestesiol. 2006 Apr;56(2):147-56. doi: 10.1590/s0034-70942006000200006. Portuguese. PMID 19468561
- [Result] Germano Filho PA, Cavalcanti IL, Barrucand L, Vercosa N. Effect of magnesium sulphate on sugammadex reversal time for neuromuscular blockade: a randomised controlled study. Anaesthesia. 2015 Aug;70(8):956-61. doi: 10.1111/anae.12987. Epub 2015 Apr 1. PMID 25829048
- [Derived] Paula-Garcia WN, Oliveira-Paula GH, de Boer HD, Garcia LV. Lidocaine combined with magnesium sulfate preserved hemodynamic stability during general anesthesia without prolonging neuromuscular blockade: a randomized, double-blind, controlled trial. BMC Anesthesiol. 2021 Mar 27;21(1):91. doi: 10.1186/s12871-021-01311-y. PMID 33773580

RESULTS

PARTICIPANT FLOW:
Recruitment Details: After approval by the Research Ethics Committee, 48 patients were selected for the study. Patients were invited to participate in the study during the pre-anesthetic evaluation, at which were told about the objectives, benefits and risks of research and those who agreed to participate signed the free consent form.
Groups:
- Group M (Magnesium Sulfate): This group received Magnesium Sulfate (MS) 40 mg/kg as a bolus over 5 minutes, followed by continuous intravenous infusion of MS 20 mg/kg/h during the surgery.
- Group ML (Magnesium Sulfate Plus Lidocaine): This group received Magnesium Sulfate (MS) 40 mg/kg plus lidocaine 3 mg/kg as a bolus over 5 minutes, followed by continuous intravenous infusion of MS 20 mg/kg/h plus lidocaine 3 mg/kg/h during the surgery.
- Group C (Control Group - Isotonic Solution): This group received isotonic solution in a equivalent volume as a bolus over 5 minutes, followed by continuous intravenous infusion of isotonic solution during the surgery.
Period: Overall Study
Arm/Group | Group M (Magnesium Sulfate) | Group ML (Magnesium Sulfate Plus Lidocaine) | Group C (Control Group - Isotonic Solution)
Started | 16 | 16 | 16
Completed | 16 | 16 | 15 (One patient required decurarization)
Not Completed | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Forty-eight 18-60 yr. old ASA I/II patients, with a body mass index of 18 - 29 kg/m2 undergoing surgery at least 90 min. were randomly allocated to 3 treatment groups.Patients who were taking medications that could affect NMB and patients with neuromuscular, renal, hepatic, cardiac dysfunction, hypermetabolic or hypometabolic states were excluded.
Groups:
- Group M: Magnesium Sulfate. In this group, the patients received magnesium sulfate 40 mg/Kg as a bolus and 20 mg/kg/h by continuous IV infusion during surgery
  Magnesium Sulfate
- Group ML: Magnesium Sulfate plus Lidocaine. In this group, the patients received 40 mg/kg of Magnesium Sulfate plus 3 mg kg-1 lidocaine as a bolus and 20 mg/kg/h and 3 mg/kg/h, respectively, by infusion continuously during the surgery
  Magnesium Sulfate
  Lidocaine
- Group C: Isotonic Solution. In this group, the patients received the volume of isotonic solution equivalent to the volume of solution infused into experimental groups
  Isotonic Solution
- Total: Total of all reporting groups
Arm/Group | Group M | Group ML | Group C | Total
Number analyzed (Participants) | 16 | 16 | 15 | 47
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 16 | 16 | 15 | 47
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 7 | 23
  Male | 8 | 8 | 8 | 24
Region of Enrollment [Number; unit: participants]
  Brazil | 16 | 16 | 15 | 47

OUTCOME MEASURES:

1. Primary Outcome: Latency
Description: The latency is computed as the elapsed time to reduce the response of T1 to 5% of the initial contraction force after the infusion of cisatracurium.
  This outcome meansure was presented in seconds.
Time Frame: Participants were followed during the anesthetic - surgical procedure, an average of 90 minutes
Population: The sample size was calculated with a power of 80% to detect differences of 20% in the timing of clinical onset and the duration of NMB. This pharmacodynamic variable was compared between the groups by analysis of variance (Anova one way) and Tukey post-hoc test (p value < 0.05)
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Group M | Group ML | Group C
Number analyzed (Participants) | 16 | 16 | 15
seconds | 139.70 (47.92) | 151.30 (47.97) | 147.80 (29.75)
Statistical Analysis 1: Comparison: Group M; Test type: Superiority or Other; p = 0.9651, ANOVA; Mean Difference (Final Values) = 149, 95% CI 2-sided [88 to 235], Standard Deviation 46.07
Statistical Analysis 2: Comparison: Group ML; Test type: Superiority or Other; p = 0.9651, ANOVA; Mean Difference (Final Values) = 145.30, 95% CI 2-sided [78 to 244], Standard Deviation 42.48
Statistical Analysis 3: Comparison: Group C; The sample size was calculated with a power of 80% to detect differences of 20% in the timing of clinical onset and the duration of NMB. The pharmacodynamic (latency, clinical duration, recovery rate and total duration) and hemodynamic variables (mean arterial pressure (MAP) and HR) were compared between the groups via analysis of variance (ANOVA) followed by the Tukey post-hoc test. The significance level was set at 5%; Test type: Superiority or Other; p = 0.9651, ANOVA; Mean Difference (Final Values) = 147.80, 95% CI 2-sided [105 to 200], Standard Deviation 29.75

2. Primary Outcome: Clinical Duration
Description: The clinical duration is the elapsed time for T1 recovery = 25% (Dur25%) of the original value of T1 after the infusion of cisatracurium.
  This outcome meansure was presented in minutes.
Time Frame: Participants were followed during the anesthetic - surgical procedure, an average of 90 minutes
Population: The sample size was calculated with a power of 80% to detect differences of 20% in the timing of clinical onset and the duration of NMB. This pharmacodynamic variable was compared between the groups by Kruskal-Wallis test. When differences were found between the groups, we used the Dunn test for multiple comparisons (p value < 0.05)
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Group M | Group ML | Group C
Number analyzed (Participants) | 16 | 16 | 15
minutes | 82.68 [76.83 to 91.19] | 86.33 [82.65 to 88.19] | 64.8 [57.05 to 70.23]
Statistical Analysis 1: Comparison: Group M; Test type: Superiority or Other; p < 0.0001, Kruskal-Wallis; Median Difference (Final Values) = 82.68, 95% CI 2-sided [72.62 to 99.27]
Statistical Analysis 2: Comparison: Group ML; Test type: Superiority or Other; p < 0.0001, Kruskal-Wallis; Median Difference (Final Values) = 86.33, 95% CI 2-sided [71.78 to 140.60]
Statistical Analysis 3: Comparison: Group C; Test type: Superiority or Other; p < 0.0001, Kruskal-Wallis; Median Difference (Final Values) = 64.80, 95% CI 2-sided [40.50 to 92.90]

3. Primary Outcome: Recovery Index
Description: The recovery index is the elapsed time between the T1 recovery =25% (Dur25%) and T1 =75% (Dur75%) after the infusion of cisatracurium.
  This outcome meansure was presented in minutes.
Time Frame: Participants were followed during the anesthetic - surgical procedure, an average of 90 minutes
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Group M | Group ML | Group C
Number analyzed (Participants) | 16 | 16 | 15
minutes | 20.08 (6.49) | 20.26 (7.69) | 14.53 (1.52)
Statistical Analysis 1: Comparison: Group M; Test type: Superiority or Other; p = 0.0015, ANOVA; Mean Difference (Final Values) = 20.08, 95% CI 2-sided [12.00 to 32.25], Standard Deviation 6.49
Statistical Analysis 2: Comparison: Group ML; Test type: Superiority or Other; p = 0.0015, ANOVA; Mean Difference (Final Values) = 20.26, 95% CI 2-sided [10.50 to 39.83], Standard Deviation 7.69
Statistical Analysis 3: Comparison: Group C; Test type: Superiority or Other; p = 0.0015, ANOVA; Mean Difference (Final Values) = 14.53, 95% CI 2-sided [11.00 to 16.50], Standard Deviation 1.52

4. Primary Outcome: Final Recovery Index
Description: The final recovery index is the elapsed time between the T1 recovery = 25% (Dur25%) and T4 / T1 = 80% (TOF = 80%) after the infusion of cisatracurium.
  This outcome measure was presented in minutes.
Time Frame: Participants were followed during the anesthetic - surgical procedure, an average of 90 minutes
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Group M | Group ML | Group C
Number analyzed (Participants) | 16 | 16 | 15
minutes | 27.97 (6.77) | 33.81 (10.97) | 21.51 (3.28)
Statistical Analysis 1: Comparison: Group M; Test type: Superiority or Other; p = 0.0003, ANOVA; Mean Difference (Final Values) = 27.97, 95% CI 2-sided [19.50 to 41.50], Standard Deviation 6.77
Statistical Analysis 2: Comparison: Group ML; Test type: Superiority or Other; p = 0.0003, ANOVA; Mean Difference (Final Values) = 33.81, 95% CI 2-sided [18.50 to 49.50], Standard Deviation 10.97
Statistical Analysis 3: Comparison: Group C; Test type: Superiority or Other; p = 0.0003, ANOVA; Mean Difference (Final Values) = 21.51, 95% CI 2-sided [17.50 to 30.05], Standard Deviation 3.28

5. Primary Outcome: Total Duration (Dur95%)
Description: The total duration is the elapsed time for T1 recovery of the response to reach 95% of the initial after the infusion of cisatracurium.
  This outcome measure was presented in minutes.
Time Frame: Participants were followed during the anesthetic - surgical procedure, an average of 90 minutes
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Group M | Group ML | Group C
Number analyzed (Participants) | 16 | 16 | 15
minutes | 113.20 (12.16) | 120.10 (18.20) | 88.19 (16.34)
Statistical Analysis 1: Comparison: Group M; Test type: Superiority or Other; p < 0.0001, ANOVA; Mean Difference (Final Values) = 113.20, 95% CI 2-sided [94.87 to 136.80], Standard Deviation 12.16
Statistical Analysis 2: Comparison: Group ML; Test type: Superiority or Other; p < 0.0001, ANOVA; Mean Difference (Final Values) = 120.10, 95% CI 2-sided [95.82 to 163.30], Standard Deviation 18.20
Statistical Analysis 3: Comparison: Group C; Test type: Superiority or Other; p < 0.0001, ANOVA; Mean Difference (Final Values) = 88.19, 95% CI 2-sided [58 to 125.20], Standard Deviation 16.34

6. Primary Outcome: Spontaneous Recovery (T4/T1=90%)
Description: Spontaneous recovery is the elapsed time for the recovery of the TOF (T4 / T1) response to 90% of the original after infusion of cisatracurium.
  This outcome measure was presented in minutes.
Time Frame: The participants were followed during the anesthetic - surgical procedure
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Group M | Group ML | Group C
Number analyzed (Participants) | 16 | 16 | 15
minutes | 120.20 (10.88) | 126.70 (14.19) | 90.03 (12.78)
Statistical Analysis 1: Comparison: Group M; Test type: Superiority or Other; p < 0.0001, ANOVA; Mean Difference (Final Values) = 120.20, 95% CI 2-sided [106.30 to 140.20], Standard Deviation 10.88
Statistical Analysis 2: Comparison: Group ML; Test type: Superiority or Other; p < 0.0001, ANOVA; Mean Difference (Final Values) = 126.70, 95% CI 2-sided [106.50 to 149.40], Standard Deviation 14.19
Statistical Analysis 3: Comparison: Group C; Test type: Superiority or Other; p < 0.0001, ANOVA; Mean Difference (Final Values) = 90.03, 95% CI 2-sided [71.75 to 116.40], Standard Deviation 12.78

7. Secondary Outcome: MAP - M1 (Mean Arterial Pressure in the Moment 1)
Description: In the operating room, patients were cardiovascular, respiratory and body temperature monitored through the Dixtal 2020. The mean blood pressure was recorded and annotated at various times such as in the arrival of the patient in the operating room. This time point was named as moment '1'.
Time Frame: This measure of average blood pressure was performed when the patient arrived in the operating room
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Group M | Group ML | Group C
Number analyzed (Participants) | 16 | 16 | 15
mmHg | 94.63 (10.18) | 88.75 (10.05) | 100.10 (16.62)
Statistical Analysis 1: Comparison: Group M; Test type: Superiority or Other; p = 0.0527, ANOVA; Mean Difference (Final Values) = 94.63, 95% CI 2-sided [70.00 to 112.00], Standard Deviation 10.18
Statistical Analysis 2: Comparison: Group ML; Test type: Superiority or Other; p = 0.0527, ANOVA; Mean Difference (Final Values) = 88.75, 95% CI 2-sided [65.00 to 104.00], Standard Deviation 10.05
Statistical Analysis 3: Comparison: Group C; Test type: Superiority or Other; p = 0.0527, ANOVA; Mean Difference (Final Values) = 100.10, 95% CI 2-sided [70.00 to 140.00], Standard Deviation 16.62

8. Secondary Outcome: MAP - M2 (Mean Arterial Pressure in the Moment 2)
Description: In the operating room, patients were cardiovascular, respiratory and body temperature monitored through the Dixtal 2020. The mean blood pressure was recorded and annotated at various times such as in the moment immediately before the anesthesia induction. This time point was named as moment '2'.
Time Frame: This measure of average blood pressure was performed immediately before induction of anesthesia
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Group M | Group ML | Group C
Number analyzed (Participants) | 16 | 16 | 15
mmHg | 87.63 (12.10) | 84.69 (11.38) | 92.47 (12.30)
Statistical Analysis 1: Comparison: Group M; Test type: Superiority or Other; p = 0.1996, ANOVA; Mean Difference (Final Values) = 87.63, 95% CI 2-sided [60.00 to 110.00], Standard Deviation 12.10
Statistical Analysis 2: Comparison: Group ML; Test type: Superiority or Other; p = 0.1996, ANOVA; Mean Difference (Final Values) = 84.69, 95% CI 2-sided [67.00 to 109.00], Standard Deviation 11.38
Statistical Analysis 3: Comparison: Group C; Test type: Superiority or Other; p = 0.1996, ANOVA; Mean Difference (Final Values) = 92.47, 95% CI 2-sided [73.00 to 112.00], Standard Deviation 12.30

9. Secondary Outcome: MAP - M3 (Mean Arterial Pressure in the Moment 3)
Description: In the operating room, patients were cardiovascular, respiratory and body temperature monitored through the Dixtal 2020. The mean blood pressure was recorded and annotated at various times such as immediately before the start of the infusion of the solution X (magnesium sulfate or isotonic solution) and Y solution (lidocaine or isotonic solution). This time point was named as moment '3'.
Time Frame: This measure of average blood pressure was performed immediately before the start of the infusion of the solution X (magnesium sulfate or isotonic solution) and Y solution (lidocaine or isotonic solution)
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Group M | Group ML | Group C
Number analyzed (Participants) | 16 | 16 | 15
mmHg | 75.88 (11.95) | 73.88 (9.80) | 76.73 (7.48)
Statistical Analysis 1: Comparison: Group M; Test type: Superiority or Other; p = 0.7145, ANOVA; Mean Difference (Final Values) = 75.88, 95% CI 2-sided [58.00 to 107.00], Standard Deviation 11.95
Statistical Analysis 2: Comparison: Group ML; Test type: Superiority or Other; p = 0.7145, ANOVA; Mean Difference (Final Values) = 73.88, 95% CI 2-sided [59.00 to 97.00], Standard Deviation 9.80
Statistical Analysis 3: Comparison: Group C; Test type: Superiority or Other; p = 0.7145, ANOVA; Mean Difference (Final Values) = 76.73, 95% CI 2-sided [58.00 to 86.00], Standard Deviation 7.48

10. Secondary Outcome: MAP - M4 (Mean Arterial Pressure in the Moment 4)
Description: In the operating room, patients were cardiovascular, respiratory and body temperature monitored through the Dixtal 2020. The mean blood pressure was recorded and annotated at various times such as in the end of the study solutions infusion.This time point was named as moment '4'.
Time Frame: This measure of average blood pressure was performed five minutes after M3 (in the end of the X and Y solutions infusion)
Measure: Median (Inter-Quartile Range); unit: mmHg
Arm/Group | Group M | Group ML | Group C
Number analyzed (Participants) | 16 | 16 | 15
mmHg | 69.00 [60.50 to 73.00] | 63.00 [60.50 to 72.00] | 74.00 [64.00 to 79.00]
Statistical Analysis 1: Comparison: Group M; Test type: Superiority or Other; p = 0.1130, Kruskal-Wallis; Median Difference (Final Values) = 69.00, 95% CI 2-sided [57.00 to 96.00]
Statistical Analysis 2: Comparison: Group ML; Test type: Superiority or Other; p = 0.1130, Kruskal-Wallis; Median Difference (Final Values) = 63.00, 95% CI 2-sided [55.00 to 84.00]
Statistical Analysis 3: Comparison: Group C; Test type: Superiority or Other; p = 0.1130, Kruskal-Wallis; Median Difference (Final Values) = 74.00, 95% CI 2-sided [59.00 to 83.00]

11. Secondary Outcome: MAP - M5 (Mean Arterial Pressure in the Moment 5)
Description: In the operating room, patients were cardiovascular, respiratory and body temperature monitored through the Dixtal 2020. The mean blood pressure was recorded and annotated at various times such as immediately before the tracheal intubation. This time point was named as moment '5'.
Time Frame: This measure of average blood pressure was performed immediately before the tracheal intubation
Measure: Median (Inter-Quartile Range); unit: mmHg
Arm/Group | Group M | Group ML | Group C
Number analyzed (Participants) | 16 | 16 | 15
mmHg | 62.50 [60.00 to 77.50] | 61.50 [57.50 to 64.25] | 67.00 [62.00 to 74.00]
Statistical Analysis 1: Comparison: Group M; Test type: Superiority or Other; p = 0.0731, Kruskal-Wallis; Median Difference (Final Values) = 62.50, 95% CI 2-sided [58.00 to 98.00]
Statistical Analysis 2: Comparison: Group ML; Test type: Superiority or Other; p = 0.0731, Kruskal-Wallis; Median Difference (Final Values) = 61.50, 95% CI 2-sided [55.00 to 74.00]
Statistical Analysis 3: Comparison: Group C; Test type: Superiority or Other; p = 0.0731, Kruskal-Wallis; Median Difference (Final Values) = 67.00, 95% CI 2-sided [56.00 to 85.00]

12. Secondary Outcome: MAP - M6 (Mean Arterial Pressure in the Moment 6)
Description: In the operating room, patients were cardiovascular, respiratory and body temperature monitored through the Dixtal 2020. The mean blood pressure was recorded and annotated at various times such as one minute after the tracheal intubation. This time point was named as moment '6'.
Time Frame: This measure of average blood pressure was performed one minute after the tracheal intubation
Measure: Median (Inter-Quartile Range); unit: mmHg
Arm/Group | Group M | Group ML | Group C
Number analyzed (Participants) | 16 | 16 | 15
mmHg | 64.50 [60.25 to 71.75] | 64.00 [60.25 to 67.75] | 69.00 [62.00 to 81.00]
Statistical Analysis 1: Comparison: Group M; Test type: Superiority or Other; p = 0.1002, Kruskal-Wallis; Median Difference (Final Values) = 64.50, 95% CI 2-sided [60.00 to 85.00]
Statistical Analysis 2: Comparison: Group ML; Test type: Superiority or Other; p = 0.1002, Kruskal-Wallis; Median Difference (Final Values) = 64.00, 95% CI 2-sided [56.00 to 74.00]
Statistical Analysis 3: Comparison: Group C; Test type: Superiority or Other; p = 0.1002, Kruskal-Wallis; Median Difference (Final Values) = 69.00, 95% CI 2-sided [60.00 to 90.00]

13. Secondary Outcome: HR - M1 (Heart Rate in the Moment 1)
Description: In the operating room, patients were cardiovascular, respiratory and body temperature monitored through the Dixtal 2020. The measure of heart rate was recorded and annotated at various times such as in the arrival of the patient in the operating room. This time point was named as moment '1'.
Time Frame: This measure of heart rate was performed when the patient arrived in the operating room
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | Group M | Group ML | Group C
Number analyzed (Participants) | 16 | 16 | 15
beats/min | 79.94 (15.79) | 77.25 (12.13) | 73.66 (11.82)
Statistical Analysis 1: Comparison: Group M; Test type: Superiority or Other; p = 0.4338, ANOVA; Mean Difference (Final Values) = 79.94, 95% CI 2-sided [52.00 to 109.00], Standard Deviation 15.79
Statistical Analysis 2: Comparison: Group ML; Test type: Superiority or Other; p = 0.4338, ANOVA; Mean Difference (Final Values) = 77.25, 95% CI 2-sided [55.00 to 95.00], Standard Deviation 12.13
Statistical Analysis 3: Comparison: Group C; Test type: Superiority or Other; p = 0.4338, ANOVA; Mean Difference (Final Values) = 73.67, 95% CI 2-sided [55.00 to 92.00], Standard Deviation 11.82

14. Secondary Outcome: HR - M2 (Heart Rate in the Moment 2)
Description: In the operating room, patients were cardiovascular, respiratory and body temperature monitored through the Dixtal 2020. The heart rate was recorded and annotated at various times such as in the moment immediately before the anesthesia induction. This time point was named as moment '2'.
Time Frame: This measure of heart rate was performed immediately before induction of anesthesia
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | Group M | Group ML | Group C
Number analyzed (Participants) | 16 | 16 | 15
beats/min | 74.69 (11.76) | 73.69 (11.18) | 75.40 (11.54)
Statistical Analysis 1: Comparison: Group M; Test type: Superiority or Other; p = 0.9167, ANOVA; Mean Difference (Final Values) = 74.69, 95% CI 2-sided [57.00 to 99.00], Standard Deviation 11.76
Statistical Analysis 2: Comparison: Group ML; Test type: Superiority or Other; p = 0.9167, ANOVA; Mean Difference (Final Values) = 73.69, 95% CI 2-sided [51.00 to 96.00], Standard Deviation 11.18
Statistical Analysis 3: Comparison: Group C; Test type: Superiority or Other; p = 0.9167, ANOVA; Mean Difference (Final Values) = 75.40, 95% CI 2-sided [53.00 to 90.00], Standard Deviation 11.54

15. Secondary Outcome: HR - M3 (Heart Rate in the Moment 3)
Description: In the operating room, patients were cardiovascular, respiratory and body temperature monitored through the Dixtal 2020. The heart rate was recorded and annotated at various times such as immediately before the start of the infusion of the solution X (magnesium sulfate or isotonic solution) and Y solution (lidocaine or isotonic solution). This time point was named as moment '3'.
Time Frame: This measure of heart rate was performed immediately before the start of the infusion of the solution X (magnesium sulfate or isotonic solution) and Y solution (lidocaine or isotonic solution)
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | Group M | Group ML | Group C
Number analyzed (Participants) | 16 | 16 | 15
beats/min | 72.94 (10.96) | 74.19 (8.65) | 75.40 (11.54)
Statistical Analysis 1: Comparison: Group M; Test type: Superiority or Other; p = 0.8067, ANOVA; Mean Difference (Final Values) = 72.94, 95% CI 2-sided [58.00 to 92.00], Standard Deviation 10.96
Statistical Analysis 2: Comparison: Group ML; Test type: Superiority or Other; p = 0.8067, ANOVA; Mean Difference (Final Values) = 74.19, 95% CI 2-sided [57.00 to 86.00], Standard Deviation 8.65
Statistical Analysis 3: Comparison: Group C; Test type: Superiority or Other; p = 0.8067, ANOVA; Mean Difference (Final Values) = 75.40, 95% CI 2-sided [53.00 to 90.00], Standard Deviation 11.54

16. Secondary Outcome: HR - M4 (Heart Rate in the Moment 4)
Description: In the operating room, patients were cardiovascular, respiratory and body temperature monitored through the Dixtal 2020. The heart rate was recorded and annotated at various times such as in the end of the study solutions infusion. This time point was named as moment '4'.
Time Frame: This measure of heart rate was performed five minutes after M3 (in the end of the X and Y solutions infusion)
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | Group M | Group ML | Group C
Number analyzed (Participants) | 16 | 16 | 15
beats/min | 71.94 (10.87) | 72.25 (9.78) | 65.07 (10.01)
Statistical Analysis 1: Comparison: Group M; Test type: Superiority or Other; p = 0.1015, ANOVA; Mean Difference (Final Values) = 71.94, 95% CI 2-sided [57.00 to 93.00], Standard Deviation 10.87
Statistical Analysis 2: Comparison: Group ML; Test type: Superiority or Other; p = 0.1015, ANOVA; Mean Difference (Final Values) = 72.25, 95% CI 2-sided [52.00 to 89.00], Standard Deviation 9.78
Statistical Analysis 3: Comparison: Group C; Test type: Superiority or Other; p = 0.1015, ANOVA; Mean Difference (Final Values) = 65.07, 95% CI 2-sided [44.00 to 81.00], Standard Deviation 10.01

17. Secondary Outcome: HR - M5 (Heart Rate in the Moment 5)
Description: In the operating room, patients were cardiovascular, respiratory and body temperature monitored through the Dixtal 2020. The heart rate was recorded and annotated at various times such as immediately before the tracheal intubation. This time point was named as moment '5'.
Time Frame: This measure of heart rate was performed immediately before the tracheal intubation
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | Group M | Group ML | Group C
Number analyzed (Participants) | 16 | 16 | 15
beats/min | 67.56 (10.05) | 69.31 (7.73) | 64.27 (10.81)
Statistical Analysis 1: Comparison: Group M; Test type: Superiority or Other; p = 0.3423, ANOVA; Mean Difference (Final Values) = 67.56, 95% CI 2-sided [56.00 to 92.00], Standard Deviation 10.05
Statistical Analysis 2: Comparison: Group ML; Test type: Superiority or Other; p = 0.3423, ANOVA; Mean Difference (Final Values) = 69.31, 95% CI 2-sided [57.00 to 83.00], Standard Deviation 7.73
Statistical Analysis 3: Comparison: Group C; Test type: Superiority or Other; p = 0.3423, ANOVA; Mean Difference (Final Values) = 64.27, 95% CI 2-sided [41.00 to 81.00], Standard Deviation 10.81

18. Secondary Outcome: HR - M6 (Heart Rate in the Moment 6)
Description: In the operating room, patients were cardiovascular, respiratory and body temperature monitored through the Dixtal 2020. The heart rate was recorded and annotated at various times such as one minute after the tracheal intubation. This time point was named as moment '6'.
Time Frame: This measure of heart rate was performed one minute after the tracheal intubation
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | Group M | Group ML | Group C
Number analyzed (Participants) | 16 | 16 | 15
beats/min | 66.50 (10.11) | 68.19 (8.40) | 65.13 (10.50)
Statistical Analysis 1: Comparison: Group M; Test type: Superiority or Other; p = 0.6817, ANOVA; Mean Difference (Final Values) = 66.50, 95% CI 2-sided [53.00 to 92.00], Standard Deviation 10.11
Statistical Analysis 2: Comparison: Group ML; Test type: Superiority or Other; p = 0.6817, ANOVA; Mean Difference (Final Values) = 68.19, 95% CI 2-sided [54.00 to 82.00], Standard Deviation 8.40
Statistical Analysis 3: Comparison: Group C; Test type: Superiority or Other; p = 0.6817, ANOVA; Mean Difference (Final Values) = 65.13, 95% CI 2-sided [47.00 to 81.00], Standard Deviation 10.50

19. Secondary Outcome: MAP - M7a (Mean Arterial Pressure in the Moment 7a)
Description: In the operating room, patients were cardiovascular, respiratory and body temperature monitored through the Dixtal 2020. The mean blood pressure was recorded and annotated at various times such as 15 minutes after the traqueal intubation. This time point was named as moment '7a'.
Time Frame: This measure of average blood pressure was performed 15 minutes after the traqueal intubation
Measure: Median (Inter-Quartile Range); unit: mmHg
Arm/Group | Group M | Group ML | Group C
Number analyzed (Participants) | 16 | 16 | 15
mmHg | 66.00 [60.75 to 73.00] | 61.50 [60.00 to 67.75] | 69.00 [63.00 to 79.00]
Statistical Analysis 1: Comparison: Group M; Test type: Superiority or Other; p = 0.0937, Kruskal-Wallis; Median Difference (Final Values) = 66.00, 95% CI 2-sided [58.00 to 80.00]
Statistical Analysis 2: Comparison: Group ML; Test type: Superiority or Other; p = 0.0937, Kruskal-Wallis; Median Difference (Final Values) = 61.50, 95% CI 2-sided [56.00 to 90.00]
Statistical Analysis 3: Comparison: Group C; Test type: Superiority or Other; p = 0.0937, Kruskal-Wallis; Median Difference (Final Values) = 69.00, 95% CI 2-sided [58.00 to 87.00]

20. Secondary Outcome: MAP - M7b (Mean Arterial Pressure in the Moment 7b)
Description: In the operating room, patients were cardiovascular, respiratory and body temperature monitored through the Dixtal 2020. The mean blood pressure was recorded and annotated at various times such as 30 minutes after the traqueal intubation. This time point was named as moment '7b'.
Time Frame: This measure of average blood pressure was performed 30 minutes after the traqueal intubation
Measure: Median (Inter-Quartile Range); unit: mmHg
Arm/Group | Group M | Group ML | Group C
Number analyzed (Participants) | 16 | 16 | 15
mmHg | 66.50 [64.25 to 74.00] | 63.50 [57.50 to 72.00] | 68.00 [62.00 to 77.00]
Statistical Analysis 1: Comparison: Group M; Test type: Superiority or Other; p = 0.1406, Kruskal-Wallis; Median Difference (Final Values) = 66.50, 95% CI 2-sided [60.00 to 88.00]
Statistical Analysis 2: Comparison: Group ML; Test type: Superiority or Other; p = 0.1406, Kruskal-Wallis; Median Difference (Final Values) = 63.50, 95% CI 2-sided [55.00 to 86.00]
Statistical Analysis 3: Comparison: Group C; Test type: Superiority or Other; p = 0.1406, Kruskal-Wallis; Median Difference (Final Values) = 68.00, 95% CI 2-sided [55.00 to 84.00]

21. Secondary Outcome: MAP - M7c (Mean Arterial Pressure in the Moment 7c)
Description: In the operating room, patients were cardiovascular, respiratory and body temperature monitored through the Dixtal 2020. The mean blood pressure was recorded and annotated at various times such as 45 minutes after the traqueal intubation. This time point was named as moment '7c'.
Time Frame: This measure of average blood pressure was performed 45 minutes after the traqueal intubation
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Group M | Group ML | Group C
Number analyzed (Participants) | 16 | 16 | 15
mmHg | 69.25 (6.74) | 63.00 (7.62) | 69.00 (7.56)
Statistical Analysis 1: Comparison: Group M; Test type: Superiority or Other; p = 0.0504, ANOVA; Mean Difference (Final Values) = 69.25, 95% CI 2-sided [60.00 to 81.00], Standard Deviation 6.74
Statistical Analysis 2: Comparison: Group ML; Test type: Superiority or Other; p = 0.0504, ANOVA; Mean Difference (Final Values) = 63.00, 95% CI 2-sided [49.00 to 79.00], Standard Deviation 7.62
Statistical Analysis 3: Comparison: Group C; Test type: Superiority or Other; p = 0.0504, ANOVA; Mean Difference (Final Values) = 69.00, 95% CI 2-sided [58.00 to 84.00], Standard Deviation 7.56

22. Secondary Outcome: MAP - M7d (Mean Arterial Pressure in the Moment 7d)
Description: In the operating room, patients were cardiovascular, respiratory and body temperature monitored through the Dixtal 2020. The mean blood pressure was recorded and annotated at various times such as 60 minutes after the traqueal intubation. This time point was named as moment '7d'.
Time Frame: This measure of average blood pressure was performed 60 minutes after the traqueal intubation
Measure: Median (Inter-Quartile Range); unit: mmHg
Arm/Group | Group M | Group ML | Group C
Number analyzed (Participants) | 16 | 16 | 15
mmHg | 68.00 [66.00 to 78.00] | 62.00 [58.25 to 69.50] | 66.00 [63.00 to 71.00]
Statistical Analysis 1: Comparison: Group M; Test type: Superiority or Other; p = 0.0205, Kruskal-Wallis; Median Difference (Final Values) = 68.00, 95% CI 2-sided [60.00 to 93.00]
Statistical Analysis 2: Comparison: Group ML; Test type: Superiority or Other; p = 0.0205, Kruskal-Wallis; Median Difference (Final Values) = 62.00, 95% CI 2-sided [54.00 to 72.00]
Statistical Analysis 3: Comparison: Group C; Test type: Superiority or Other; p = 0.0205, Kruskal-Wallis; Median Difference (Final Values) = 66.00, 95% CI 2-sided [59.00 to 75.00]

23. Secondary Outcome: MAP - M7e (Mean Arterial Pressure in the Moment 7e)
Description: In the operating room, patients were cardiovascular, respiratory and body temperature monitored through the Dixtal 2020. The mean blood pressure was recorded and annotated at various times such as 75 minutes after the traqueal intubation. This time point was named as moment '7e'.
Time Frame: This measure of average blood pressure was performed 75 minutes after the traqueal intubation
Measure: Median (Inter-Quartile Range); unit: mmHg
Arm/Group | Group M | Group ML | Group C
Number analyzed (Participants) | 16 | 16 | 15
mmHg | 68.00 [61.25 to 76.50] | 66.00 [59.00 to 69.75] | 69.00 [65.00 to 73.00]
Statistical Analysis 1: Comparison: Group M; Test type: Superiority or Other; p = 0.3004, Kruskal-Wallis; Median Difference (Final Values) = 68.00, 95% CI 2-sided [58.00 to 86.00]
Statistical Analysis 2: Comparison: Group ML; Test type: Superiority or Other; p = 0.3004, Kruskal-Wallis; Median Difference (Final Values) = 66.00, 95% CI 2-sided [56.00 to 78.00]
Statistical Analysis 3: Comparison: Group C; Test type: Superiority or Other; p = 0.3004, Kruskal-Wallis; Median Difference (Final Values) = 69.00, 95% CI 2-sided [62.00 to 81.00]

24. Secondary Outcome: MAP - M7f (Mean Arterial Pressure in the Moment 7f)
Description: In the operating room, patients were cardiovascular, respiratory and body temperature monitored through the Dixtal 2020. The mean blood pressure was recorded and annotated at various times such as 90 minutes after the traqueal intubation. This time point was named as moment '7f'.
Time Frame: This measure of average blood pressure was performed 90 minutes after the traqueal intubation
Measure: Median (Inter-Quartile Range); unit: mmHg
Arm/Group | Group M | Group ML | Group C
Number analyzed (Participants) | 16 | 16 | 15
mmHg | 64.00 [62.00 to 77.00] | 64.50 [60.00 to 70.00] | 72.00 [68.00 to 80.00]
Statistical Analysis 1: Comparison: Group M; Test type: Superiority or Other; p = 0.0178, Kruskal-Wallis; Median Difference (Final Values) = 64.00, 95% CI 2-sided [60.00 to 84.00]
Statistical Analysis 2: Comparison: Group ML; Test type: Superiority or Other; p = 0.0178, Kruskal-Wallis; Median Difference (Final Values) = 64.50, 95% CI 2-sided [51.00 to 75.00]
Statistical Analysis 3: Comparison: Group C; Test type: Superiority or Other; p = 0.0178, Kruskal-Wallis; Median Difference (Final Values) = 72.00, 95% CI 2-sided [61.00 to 91.00]

25. Secondary Outcome: HR - M7a (Heart Rate in the Moment 7a)
Description: In the operating room, patients were cardiovascular, respiratory and body temperature monitored through the Dixtal 2020. The heart rate was recorded and annotated at various times such as 15 minutes after the traqueal intubation.This time point was named as moment '7a'.
Time Frame: This measure of heart rate was performed 15 minutes after the traqueal intubation
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | Group M | Group ML | Group C
Number analyzed (Participants) | 16 | 16 | 15
beats/min | 68.94 (11.99) | 68.19 (7.73) | 67.13 (8.85)
Statistical Analysis 1: Comparison: Group M; Test type: Superiority or Other; p = 0.8746, ANOVA; Mean Difference (Final Values) = 68.67, 95% CI 2-sided [51.00 to 99.00], Standard Deviation 8.51
Statistical Analysis 2: Comparison: Group ML; Test type: Superiority or Other; p = 0.8746, ANOVA; Mean Difference (Final Values) = 64.38, 95% CI 2-sided [56.00 to 82.00], Standard Deviation 6.96
Statistical Analysis 3: Comparison: Group C; Test type: Superiority or Other; p = 0.8746, ANOVA; Mean Difference (Final Values) = 73.40, 95% CI 2-sided [54.00 to 80.00], Standard Deviation 7.94

26. Secondary Outcome: HR - M7b (Heart Rate in the Moment 7b)
Description: In the operating room, patients were cardiovascular, respiratory and body temperature monitored through the Dixtal 2020. The heart rate was recorded and annotated at various times such as 30 minutes after the traqueal intubation. This time point was named as moment '7b'.
Time Frame: This measure of heart rate was performed 30 minutes after the traqueal intubation
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | Group M | Group ML | Group C
Number analyzed (Participants) | 16 | 16 | 15
beats/min | 67.44 (10.95) | 68.38 (9.28) | 64.00 (8.23)
Statistical Analysis 1: Comparison: Group M; Test type: Superiority or Other; p = 0.4195, ANOVA; Mean Difference (Final Values) = 67.44, 95% CI 2-sided [47.00 to 92.00], Standard Deviation 10.95
Statistical Analysis 2: Comparison: Group ML; Test type: Superiority or Other; p = 0.4195, ANOVA; Mean Difference (Final Values) = 68.38, 95% CI 2-sided [53.00 to 80.00], Standard Deviation 9.28
Statistical Analysis 3: Comparison: Group C; Test type: Superiority or Other; p = 0.4195, ANOVA; Mean Difference (Final Values) = 64.00, 95% CI 2-sided [52.00 to 80.00], Standard Deviation 8.23

27. Secondary Outcome: HR - M7c (Heart Rate in the Moment 7c)
Description: In the operating room, patients were cardiovascular, respiratory and body temperature monitored through the Dixtal 2020. The heart rate was recorded and annotated at various times such as 45 minutes after the traqueal intubation. This time point was named as moment '7c'.
Time Frame: This measure of heart rate was performed 45 minutes after the traqueal intubation
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | Group M | Group ML | Group C
Number analyzed (Participants) | 16 | 16 | 15
beats/min | 65.75 (11.52) | 65.75 (10.19) | 62.33 (9.26)
Statistical Analysis 1: Comparison: Group M; Test type: Superiority or Other; p = 0.5796, ANOVA; Mean Difference (Final Values) = 65.75, 95% CI 2-sided [47.00 to 93.00], Standard Deviation 11.52
Statistical Analysis 2: Comparison: Group ML; Test type: Superiority or Other; p = 0.5796, ANOVA; Mean Difference (Final Values) = 65.75, 95% CI 2-sided [48.00 to 79.00], Standard Deviation 10.19
Statistical Analysis 3: Comparison: Group C; Test type: Superiority or Other; p = 0.5796, ANOVA; Mean Difference (Final Values) = 62.33, 95% CI 2-sided [50.00 to 79.00], Standard Deviation 9.26

28. Secondary Outcome: HR - M7d (Heart Rate in the Moment 7d)
Description: In the operating room, patients were cardiovascular, respiratory and body temperature monitored through the Dixtal 2020. The heart rate was recorded and annotated at various times such as 60 minutes after the traqueal intubation. This time point was named as moment '7d'.
Time Frame: This measure of heart rate was performed 60 minutes after the traqueal intubation
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | Group M | Group ML | Group C
Number analyzed (Participants) | 16 | 16 | 15
beats/min | 66.19 (12.82) | 65.31 (10.87) | 61.93 (9.00)
Statistical Analysis 1: Comparison: Group M; Test type: Superiority or Other; p = 0.5351, ANOVA; Mean Difference (Final Values) = 66.19, 95% CI 2-sided [45.00 to 92.00], Standard Deviation 12.82
Statistical Analysis 2: Comparison: Group ML; Test type: Superiority or Other; p = 0.5351, ANOVA; Mean Difference (Final Values) = 65.31, 95% CI 2-sided [47.00 to 82.00], Standard Deviation 10.87
Statistical Analysis 3: Comparison: Group C; Test type: Superiority or Other; p = 0.5351, ANOVA; Mean Difference (Final Values) = 61.93, 95% CI 2-sided [51.00 to 79.00], Standard Deviation 9.00

29. Secondary Outcome: HR - M7e (Heart Rate in the Moment 7e)
Description: In the operating room, patients were cardiovascular, respiratory and body temperature monitored through the Dixtal 2020. The heart rate was recorded and annotated at various times such as 75 minutes after the traqueal intubation. This time point was named as moment '7e'.
Time Frame: This measure of heart rate was performed 75 minutes after the traqueal intubation
Measure: Median (Inter-Quartile Range); unit: beats/min
Arm/Group | Group M | Group ML | Group C
Number analyzed (Participants) | 16 | 16 | 15
beats/min | 66.50 [54.00 to 71.75] | 63.00 [56.00 to 72.75] | 58.00 [54.00 to 65.00]
Statistical Analysis 1: Comparison: Group M; Test type: Superiority or Other; p = 0.4988, Kruskal-Wallis; Median Difference (Final Values) = 66.50, 95% CI 2-sided [42.00 to 92.00]
Statistical Analysis 2: Comparison: Group ML; Test type: Superiority or Other; p = 0.4988, Kruskal-Wallis; Median Difference (Final Values) = 63.00, 95% CI 2-sided [50.00 to 85.00]
Statistical Analysis 3: Comparison: Group C; Test type: Superiority or Other; p = 0.4988, Kruskal-Wallis; Median Difference (Final Values) = 58.00, 95% CI 2-sided [51.00 to 80.00]

30. Secondary Outcome: HR - M7f (Heart Rate in the Moment 7f)
Description: In the operating room, patients were cardiovascular, respiratory and body temperature monitored through the Dixtal 2020. The heart rate was recorded and annotated at various times such as 90 minutes after the traqueal intubation. This time point was named as moment '7f'.
Time Frame: This measure of heart rate was performed 90 minutes after the traqueal intubation
Measure: Median (Inter-Quartile Range); unit: beats/min
Arm/Group | Group M | Group ML | Group C
Number analyzed (Participants) | 16 | 16 | 15
beats/min | 66.00 [53.50 to 70.00] | 61.00 [55.00 to 64.00] | 61.00 [55.75 to 73.75]
Statistical Analysis 1: Comparison: Group M; Test type: Superiority or Other; p = 0.7723, Kruskal-Wallis; Median Difference (Final Values) = 66.00, 95% CI 2-sided [43.00 to 89.00]
Statistical Analysis 2: Comparison: Group ML; Test type: Superiority or Other; p = 0.7723, Kruskal-Wallis; Median Difference (Final Values) = 61.00, 95% CI 2-sided [51.00 to 82.00]
Statistical Analysis 3: Comparison: Group C; Test type: Superiority or Other; p = 0.7723, Kruskal-Wallis; Median Difference (Final Values) = 61.00, 95% CI 2-sided [50.00 to 78.00]

ADVERSE EVENTS:
Time Frame: The adverse event data were collected during the intra and posopertive period.
Arm/Group | Group M | Group ML | Group C
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16 | 0/15
Other Adverse Events (participants affected / at risk) | 0/16 | 0/16 | 0/15

LIMITATIONS AND CAVEATS:
-It was not possible to measure Magnesium sulfate and Lidocaine levels

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No